CLINICAL TRIAL: NCT03315793
Title: A Double-blind, Efficacy and Safety Study of Duloxetine Hydrochloride Versus Placebo in the Treatment of Japanese Children and Adolescents With Depressive Disorder
Brief Title: A Study of Duloxetine (LY248686) in Japanese Children and Adolescents With Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14937; F1J-JE-B058 (Other: Eli Lilly and Company); 1701A3631 (Other: Shionogi)
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12-01

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Duloxetine Hydrochloride (Experimental): Duloxetine hydrochloride given orally.
  Interventions: Drug: Duloxetine Hydrochloride
- Placebo (Placebo Comparator): Placebo given orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine Hydrochloride — Administered orally
  Other Names: LY248686
  Arms: Duloxetine Hydrochloride
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of duloxetine hydrochloride versus placebo in the treatment of Japanese children and adolescents with depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with Major Depressive Disorder or persistent depressive disorder and completely meet the criteria of major depressive episode as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) with the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) ver.7.0.2.
* Participants whose incipient age of depression was ≥7 years old.
* Total score of CDRS-R is ≥40 and CGI-S score is ≥4 at both screening and baseline.

Exclusion Criteria:

* Have remarkable response to psycho-education (defined as >30% decrease in the total score of CDRS-R between screening and baseline).
* Have a current or previous diagnosis (DSM-5) of the following as judged by the investigator:

  * Neurodevelopmental disorders
  * Schizophrenia spectrum and other psychotic disorders
  * Bipolar and related disorders
  * Trauma and stressor-related disorders
  * Disruptive · Impulse Control · and Conduct disorders
* Have a current diagnosis (DSM-5) of the following as judged by the investigator:

  * Obsessive-compulsive and related disorders
  * Anorexia nervosa, Bulimia nervosa, Binge-eating disorder
  * Sleep-wake disorders
  * Neurocognitive disorders
  * Disruptive mood dysregulation disorder
* Have personality disorders, in the judgement of the investigator.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trial Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (1):
- Shionogi, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Duloxetine: 20 mg Duloxetine was administered every day for 1 week. Then 40 mg Duloxetine was administered for 1 week. Then flexible doses of 40 mg or 60 mg Duloxetine were administered for 4 weeks. Lower doses of Duloxetine were administered for 1 week during tapering off period.
- Placebo: Placebo was administered every day for 7 weeks.
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 75 | 74
Received at Least 1 Dose of Study Drug | 75 | 74
Completed | 70 | 71
Not Completed | 5 | 3
Not completed — Adverse Event | 4 | 2
Not completed — Protocol Deviation | 1 | 0
Not completed — Difficult for regular visit | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of drug and had at least 1 post-dose CDRS-R Total Score. One participant in the duloxetine group had no post-dose CDRS-R Total Score and was not included in the analysis.
Groups:
- Duloxetine: 20 mg Duloxetine was administered for 1 week. Then 40 mg Duloxetine was administered for 1 week. Then flexible doses of 40 mg or 60 mg Duloxetine were administered for 4 weeks. Lower doses Duloxetine were administered for 1 week during tapering off period.
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (1.9) | 14.6 (2.0) | 14.5 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 93
  Male | 28 | 27 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 74 | 74 | 148
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 74 | 74 | 148
Children's Depression Rating Scale-Revised (CDRS-R) Total Score [Mean (Standard Deviation); unit: units on a scale] — Children's Depression Rating Scale-Revised (CDRS-R) Total score measures the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. A rating of 1 indicates normal functioning and higher numbers indicate a higher degree of depression. The total sum of scores range from 17 to 113. In general, scores below 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, scores of 40 to 60 indicate moderate depression, and scores greater than 60 indicate severe depression.
  units on a scale | 65.7 (10.5) | 63.3 (12.4) | 64.5 (11.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Children's Depression Rating Scale-Revised (CDRS-R) Total Score
Description: Change from baseline on the Children's Depression Rating Scale-Revised (CDRS-R) total score. CDRS-R Total score measures the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. A rating of 1 indicates normal functioning and a higher number indicates a greater degree of depression. The total sum of scores range from 17 to 113. In general, scores below 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, scores of 40 to 60 indicate moderate depression, and scores greater than 60 indicate severe depression. Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach including treatment group, observation time-points, and interaction between treatment group and observation time-points as fixed effects, and baseline CDRS-R total score and age as covariates.
Time Frame: Baseline, Week 6
Population: All randomized participants who received 1 dose of study drug and had 1 post-baseline CDRS-S score. One participant in the duloxetine group had no post-dose CDRS-R Total Score and was not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 74 | 74
units on a scale | -21.03 (2.04) | -22.42 (2.05)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority; p = 0.5587, mixed-effects model repeated measures; Least squares mean difference = 1.39, 98% CI 2-sided [-3.30 to 6.08]

2. Secondary Outcome: Percentage of Participants Whose Children's Depression Rating Scale-Revised (CDRS-R) Total Score Decreased by More Than 30% From Baseline
Description: The Children's Depression Rating Scale-Revised (CDRS-R) Total score measures the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. A rating of 1 indicates normal functioning and higher numbers indicate a greater degree of depression. The total sum of scores range from 17 to 113. In general, scores below 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, scores of 40 to 60 indicate moderate depression, and scores greater than 60 indicate severe depression.
Time Frame: Baseline, Week 6
Population: All randomized participants who received at least one dose of study drug and had at least 1 post-dose CDRS-R Total Score. One participant in the duloxetine group had no post-dose CDRS-R Total Score and was not included in the analysis. The last observation carried forward (LOCF) method was used.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 74 | 74
percentage of participants | 48.6 | 43.2
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority; p = 0.5111, Cochran-Mantel-Haenszel; Stratified by age; Risk Difference (RD) = 5.4, 95% CI 2-sided [-10.7 to 21.5]

3. Secondary Outcome: Percentage of Participants Whose CDRS-R Total Score Decreased by More Than 50% From Baseline
Description: The Children's Depression Rating Scale-Revised (CDRS-R) total score measures the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. A rating of 1 indicates normal functioning with higher numbers indicating a greater degree of depression . The total sum of scores range from 17 to 113. The total sum of scores range from 17 to 113. In general, scores below 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, scores of 40 to 60 indicate moderate depression, and scores greater than 60 indicate severe depression.
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 74 | 74
percentage of participants | 21.6 | 21.6
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Stratified by age; Risk Difference (RD) = 0.0, 95% CI 2-sided [-13.5 to 13.5]

4. Secondary Outcome: Percentage of Participants With Total Children's Depression Rating Scale-Revised (CDRS-R) Score ≤ 28
Description: The Children's Depression Rating Scale-Revised (CDRS-R) total score measures the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. A rating of 1 indicates normal functioning and higher numbers indicate a greater degree of depression. The total sum of scores range from 17 to 113. In general, scores below 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, scores of 40 to 60 indicate moderate depression, and scores greater than 60 indicate severe depression. Remission was defined for the CDRS-R total score below 28.
Time Frame: Baseline, Week 6
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose CDRS-R Total Score. One participant in the duloxetine group had no post-dose CDRS-R Total Score and was not included in the analysis. The last observation carried forward (LOCF) method was used.
Measure: Number; unit: percentage of participants
Groups:
- Duloxetine: 20 mg Duloxetine was administered for 1 week. Then 40 mg Duloxetine was administered for 1 week. Then flexible doses of 40 mg or 60 mg Duloxetine were administered for 4 weeks. Lower doses of Duloxetine were administered for 1 week during tapering off period.
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 74 | 74
percentage of participants | 9.5 | 13.5
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority; p = 0.4423, Cochran-Mantel-Haenszel; Stratified by age; Risk Difference (RD) = -4.1, 95% CI 2-sided [-14.4 to 6.3]

5. Secondary Outcome: Change From Baseline on Clinical Global Impression-Severity (CGI-S)
Description: CGI-S measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). Presented here are the LS mean change from baseline on CGI-S calculated using a mixed-effects model repeated measures (MMRM) approach including treatment group, observation time-points, and interaction between treatment group and observation time-points as fixed effects, and baseline CGI-S and age as covariates.
Time Frame: Baseline, Week 6
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose CDRS-R Total score. One duloxetine participant had no post-dose CDRS-R Total Score and was not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 74 | 74
units on a scale | -1.24 (0.14) | -1.38 (0.14)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority; p = 0.3836, mixed-effects model repeated measures; Least squares mean difference = 0.14, 95% CI 2-sided [-0.18 to 0.46]

ADVERSE EVENTS:
Time Frame: Baseline to 7 Weeks
Description: All participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Duloxetine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/74
Other Adverse Events (participants affected / at risk) | 59/75 | 46/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Duloxetine (N=75) | Placebo (N=74)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 2 (2)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 19 (20) | 9 (10)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 5 (5) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Thirst (General disorders) | 2 (2) | 0 (0)
Vaccination site swelling (General disorders) | 0 (0) | 1 (1)
Withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 10 (10) | 12 (12)
Otitis externa (Infections and infestations) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 2 (2) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 13 (13) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 8 (9)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 17 (17) | 8 (8)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Euphoric mood (Psychiatric disorders) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 3 (5) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 2 (2)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1/29 (1) | 0/27 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0/46 (0) | 1/47 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Yawning (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria thermal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT03315793/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT03315793/SAP_001.pdf